CLINICAL TRIAL: NCT02102308
Title: A Multicomponent Exercise Improves Executive Function and Dual-task Decrements in Gait Among Older Adults
Brief Title: Exercise Improves Executive Function and Dual-task Decrements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: elderly1; NSC100-2314-B-010-021-MY2 (Other Grant/Funding Number: NSC100-2314-B-010-021-MY2)
Record Dates: First submitted 2014-03-26; First posted 2014-04-02 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-03

CONDITIONS: Older Adults
MeSH Terms: interventions — Exercise; Prenatal Education

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise (Experimental): Multicomponent exercise
  Interventions: Other: Exercise
- Education classes (Placebo Comparator): Education classes
  Interventions: Other: Education classes

INTERVENTIONS:
Other: Exercise — Multicomponent exercise
  Arms: Exercise
Other: Education classes
  Arms: Education classes

SUMMARY:
A 12-week multicomponent exercise is effective in improving executive function and gait performance in dual-task conditions.

ELIGIBILITY:
Inclusion Criteria:

* age more than 65 years old
* ability to walk outdoor independently without assistive devices

Exclusion Criteria:

* unstable medical conditions interfering with participation in the study
* diagnosis of dementia, psychosis, neurological disease, and depression
* unable to receive external information for finishing the neuropsychological tests

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
spatial and temporal gait parameters | 12 weeks
  velocity (cm/s), stride time (ms), stride length (cm), stride time variability (%) and stride length variability (%) under single- or two dual-task conditions

SECONDARY OUTCOMES:
Executive Interview | 12 weeks
  This test consisted of 25-item rating for executive function on tasks. Scores ranged from 0 to 2 for each item, and higher scores indicated worse performance.

CONTACTS AND LOCATIONS:
Overall Officials: Yea-Ru Yang, PhD, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- Department of Physical Therapy and Assistive Technology, Taipei, Taiwan